CLINICAL TRIAL: NCT02138357
Title: Butrans for Treatment of Restless Legs Syndrome
Acronym: Butrans
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Winkelman, MD, PhD, Chief of the Sleep Disorders Clinical Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013D004946
Record Dates: First submitted 2014-05-09; First posted 2014-05-14 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Willis Ekbom Disease; Twitchy Legs; Periodic Limb Movements; Leg Movements; Augmentation; Requip; ropinirole; Mirapex; pramipexole; gabapentin; Horizant; Neupro; rotigotine
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Patch (Placebo Comparator): The Placebo is in the form of a patch. We will be using placebo patches labeled 5mcg/hour, 10mcg/hour, and 20mcg/hour that will be changed every 7 days.
  Each subject will participate in this arm of the study for four weeks.
  Interventions: Drug: buprenorphine transdermal delivery system (BTDS); Drug: Placebo for BTDS patch
- buprenorphine transdermal delivery system (BTDS) (Experimental): buprenorphine transdermal delivery system (BTDS), brand name Butrans. Butrans is in the form of a patch. We will be using 5mcg/hour, 10mcg/hour, and 20mcg/hour patches that will be changed every 7 days.
  Each subject will participate in this arm of the study for four weeks.
  Interventions: Drug: buprenorphine transdermal delivery system (BTDS); Drug: Placebo for BTDS patch

INTERVENTIONS:
Drug: buprenorphine transdermal delivery system (BTDS)
  Other Names: Butrans
Drug: Placebo for BTDS patch — A placebo patch will be manufactured to mimic the BTDS patch.

SUMMARY:
The primary objective of the study is to determine whether Butrans Transdermal System (BTDS) reduces RLS symptom severity in patients with moderate to severe idiopathic RLS who are naïve to opiate treatment.

The secondary objective of the study is to investigate the effects of BTDS on mood, sleep, and quality of life.

The study will consist of nine visits. Depending on the need for medication titration, there may also be two scheduled telephone contacts.

Visit 1: This is a screening visit to determine study eligibility. Eligible subjects who choose to participate must undergo medication washout as described in the detailed protocol between visits 1 and 2.

Treatment period #1 (Visits 2 - 5; day 0 - 28): Baseline measures will be recorded and subjects randomized to treatment order at visit 2 (day 0). Study medication as well as rescue medication (l-dopa, a non-blinded active treatment to be used within a limited dose range as described in the detailed protocol) will be dispensed. Subjects will begin treatment period #1 immediately after this. The study medication will be titrated within the allowed range according to subject's reported symptoms during visit 3 (day 7), visit 4 (day 14), telephone contact (day 21). Visit 5 will occur on day 28 and will include assessment of outcome measures for the first treatment period. Visit 5 will also mark the beginning of the second treatment period.

Treatment period #2 (Visits 6 - 8; day 28 - 56): Procedures will be similar to those described above during treatment period #1. Visit 8 will mark the end of the second treatment period during which outcome measures will be ascertained.

Follow up visit (Visit 9; day 70): This will be a safety follow-up visit approximately two weeks after visit 8 for review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of RLS, defined by International Restless Legs Study Group (IRLS) essential criteria:

  * An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs.
  * The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying down or sitting.
  * The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
  * The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night.
* Subject has moderate to severe RLS symptoms,defined as an International Restless Legs Scale (IRLS) score greater than or equal to15 at the baseline visit (visit 2).
* Subject has RLS symptoms that, in the opinion of the investigator, require round-the-clock treatment.
* Subject speaks and reads English.
* Subject is able to provide informed consent.
* Subject is age ≥25 and ≤75.
* Subject has BMI ≥18 and ≤35
* Subject is naïve to opioid treatment, defined as subjects not having received ≥5 mg oxycodone in the past 14 days and no history of daily use of ≥5 mg oxycodone equivalents in the past 3 months.
* If subject is currently being treated for RLS, s/he must have an inadequate response to or be intolerant of current, non-opioid regimen.
* If subject is not currently being treated for RLS, s/he must have a contraindication to or a history of intolerance to non-opioid treatment options for RLS, concerns about side effects of such options, or a preference for non-oral medication.
* If subject is currently being treated with a medication for RLS, a washout period of at least 3 days will be required (or 5 half-lives for longer-acting agents).
* Subject's history and/or clinical records document no change in medications active in the central nervous system (antidepressants, analgesics, antipsychotics, antiepileptics, hypnotics, etc.) for at least 30 days prior to visit 1.
* Subject is able to understand study procedures and agrees to remain on stable medications during the period of the study.
* Women of childbearing potential must agree to use a medically accepted method of birth control. Acceptable forms of birth control include:
* Condom + spermicide
* Diaphragm + spermicide
* Oral contraceptive pills, hormone implants (like Norplant), or injections(like Depo-Provera)
* Intrauterine Device

Exclusion Criteria:

* Lifetime history of DSM-IVopiod, alcohol, or other substance abuse.
* History of opioid treatment for RLS with inadequate response
* Positive urine toxicology screen at visit 1.
* Another chronic pain syndrome that would, in the opinion of the investigator, interfere with evaluation of RLS symptoms or the response to the study medication.
* Plan to undergo a procedure that may require short or long-term opiates for pain control during the course of the trial.
* History of severe mental illness.
* Women who are pregnant, lactating, or planning to become pregnant.
* Shift work or other commitments that do not allow for regular sleep at night.
* Known hypersensitivity or intolerance to opioids.
* History of Long QT Syndrome or an immediate family member with this condition, or known prolongation of QTc interval.
* QTc interval prolongation >500 ms on screening EKG at Visit 1.
* History of malignant melanoma.
* Current use of monoamine oxidase inhibitors.
* Prior or current clinically significant impulse control disorder, as determined by clinical interview and the Modified Minnesota Impulse Disorders Interview at Visit 1.8
* Untreated severe sleep apnea, defined as AHI >30.
* Iron deficiency, defined as ferritin<15 at Visit 1.
* Any dermatologic condition resulting in widespread compromise of skin integrity, defined as >50% of the surface area within the 8 sites described for BTDS application.
* Current use of class IA or class III anti-arrhythmic medication.
* Significant risk for suicide by clinical interview.
* Known hypersensitivity to buprenorphine or any excipient of BTDS.
* Current unstable medical illness.
* Any medical or psychiatric condition that, in the opinion of the investigator, would interfere with participation in the study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04 (Estimated); Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The International Restless Legs Scale (IRLS) | Within subjects IRLS score change after 4 weeks on placebo vs 4 weeks on BTDS
  The primary endpoint will be the within-subjects difference in IRLS between BTDS and placebo treatment, measured at visits 5 and 8. This comparison will be made with a fixed effects model in SAS, using PROC MIXED with a repeated statement (baseline, BTDS, placebo) to account for intra-subject correlation. Sequence, treatment, and treatment by sequence interactionterms will be included as fixed effects.

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement | Evaluated after 4 weeks on placebo and again after 4 weeks on BTDS or vice versa
  The main secondary endpoint will be the difference between placebo and BTDS in the percentage of subjects who are "much improved" or "very much improved" on the CGI-I, evaluated using generalized estimating equations.

OTHER OUTCOMES:
MOS Sleep Scales | Evaluated after 4 weeks on placebo and again after 4 weeks on BTDS or vice versa
  Another secondary endpoint will be the difference between BTDS and placebo on the MOS Sleep Scales (sleep disturbance, sleep quantity, and sleep adequacy).
Profile of Mood States (POMS) | Evaluated after 4 weeks on placebo and again after 4 weeks on BTDS or vice versa
  Another secondary endpoint will be the difference between BTDS and placebo on the Profile of Mood States (POMS).
RLS-QLI | Evaluated after 4 weeks on placebo and again after 4 weeks on BTDS or vice versa
  Another secondary endpoint will be the difference between BTDS and placebo on the RLS Quality of Life Questionnaire (RLS-QLI).

CONTACTS AND LOCATIONS:
Overall Officials: John W. Winkelman, MD, PhD, Principal Investigator — Massachusetts General Hospital (Partners Healthcare)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States